CLINICAL TRIAL: NCT00534677
Title: Efficacy And Safety Of Terlipressin Vs Octreotide As Adjuvant Therapy In Bleeding Esophageal Varices
Brief Title: The Safety & Efficacy of Terlipressin vs Octreotide for the Control of Variceal Bleed
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Dr. Shahab Abid, The Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 297-Med/ERC-04
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-09

CONDITIONS: Portal Hypertension; Cirrhosis; Hematemesis; Melena
Keywords: Variceal bleed; Cirrhosis; Vasoactive agents; Terlipressin; Octreotide; Safety & Efficacy
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; Hematemesis; Melena | interventions — Terlipressin; Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Terlipressin
- B (Active Comparator)
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Terlipressin — 2 mg stat & then 1 mg q6h iv and Placebo of Octreotide
  Other Names: Novapresin
  Arms: A
Drug: Octreotide — Octreotide 50mcg/hr infusion & a placebo of Terlipressin
  Other Names: sandostatin
  Arms: B

SUMMARY:
Terlipressin and Octreotide are two common agents used as adjuvants in the management of variceal bleeding. Both agents have been claimed equivalent to endoscopic therapy in randomized studies. There are no head to head clinical trials of these two agents available in the literature. We aimed to compare the efficacy and safety of Terlipressin and Octreotide in combination with Endoscopic Variceal band Ligation (EVL)in patients presenting with Esophageal Variceal Bleed (EVB).

DETAILED DESCRIPTION:
The effectiveness of combining Endoscopic treatment with Octreotide or Terlipressin has not been prospectively studied in esophageal variceal hemorrhage (EVH).

This prospective, randomized clinical trial will help us in better patient management more efficiently and cost effectively.

ELIGIBILITY:
Inclusion Criteria:

* All cirrhotic patients with upper GI bleed secondary to esophageal varices of 18 years or more of age

Exclusion Criteria:

* Ulcerative esophagitis,
* Mallory Weiss tear,
* Bleeding gastric or duodenal ulcers,
* Bleeding from gastric varices or portal hypertensive gastropathy and
* Upper GI bleed as a result of thrombocytopenia or bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2004-05; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Safety & Efficacy | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Abid, FCPS, FACG, Principal Investigator — Aga Khan University; Wasim Jafri, FRCP, FACG, Study Director — Aga Khan University; Saeed S Hamid, FRCP, FACG, Study Director — Aga Khan University; Salih Mohammad, FCPS; MACG, Study Director — Aga Khan University
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan